CLINICAL TRIAL: NCT01891578
Title: Evaluation of Immunological Reconstitution After Haploidentical Bone Marrow Transplantation Using a Nonmyeloablative Preparative Regimen and Post-transplant Cyclophosphamide, in Patients With Poor Prognosis Lymphomas
Brief Title: Evaluation of Immunological Reconstitution After Haploidentical Bone Marrow Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-04/2010
Record Dates: First submitted 2013-05-27; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of immunological reconstitution after haploidentical BMT using a nonmyeloablative preparative regimen and post-transplant cyclophosphamide in patients with poor prognosis lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma (any histology) relapsed after high dose chemotherapy and in partial remission, complete remission or stable disease after the last CT line that
* Signed informed consent to perform an haploidentical allo-BMT using a nonmyeloablative preparative regimen and post-transplant cyclophosphamide

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma (any histology)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of T lymphocytes and NK cells absolute number | 1 year

SECONDARY OUTCOMES:
Evaluation of discrete T-cells populations | 1 year
  Evaluation, by flow cytometry, of discrete T cell populations, including CD4+ and CD8+ TN, TSCM, TCM and TEM, NK and NKT cells, B cells, dendritic cell subsets
Evaluation of antigen-specific T cell populations | 1 year
  Evaluation of antigen-specific T cell frequency towards CMV, EBV and influenza virus by MHC tetramers
Evaluation of antigen-specific T lymphocyte's functionality | 1 year
  antigen-specific T lymphocyte's functionality towards tumor cell line evaluated using a degranulation assay
Evaluation of cytokines production by IL-2 and anti-CD16 activated NK cells | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy